CLINICAL TRIAL: NCT02127554
Title: Langzeitresultate Und Komplikationen Nach Einer Epistaxisbehandlung
Brief Title: Long Term Results and Complications After Epistaxis Treatment
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: SM_21_01_2014; KEK-ZH-Nr: 2013-0519 (Other: Zurich Ethics Committee)
Record Dates: First submitted 2014-04-28; First posted 2014-04-30 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2015-12

CONDITIONS: Nosebleed (Epistaxis) - Posterior or Anterior
MeSH Terms: conditions — Epistaxis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (7):
- Electric coagulation: Patients with anterior epistaxis, treated with electric coagulation
- Chemical coagulation: Patients with anterior epistaxis, treated with chemical coagulation
- Outpatient tamponade: Patients with posterior epistaxis, treated with tamponade as an outpatient
- Inpatient tamponade: Patients with posterior epistaxis, treated with tamponade and kept in the hospital.
- Surgery: Patients with posterior epistaxis, treated with surgery as inpatients
- Foley balloon catheter: Patients with posterior epistaxis, treated as inpatients with Foley balloon catheter
- Combined treatment: Patients with posterior epistaxis, treated as inpatients with a combination of methods

SUMMARY:
The aim of this study is to find the most agreeable and in the long term most efficient treatment for epistaxis.

DETAILED DESCRIPTION:
In the general population epistaxis occurs quite frequently. Approximately 60% of persons will be affected once in their lifetime, and 6% thereof will seek medical advice. Thereby anterior and posterior epistaxis are discerned. Anterior epistaxis is usually located at the Locus Kisselbachii, while posterior bleeds are found further back in the nose. There, most bleeds will originate from the A. sphenopalatina or the A. ethmoidalis.

Different treatment modalities exist. Anterior epistaxis are usually easier to treat than posterior ones. The aim of this study is to find the most efficient treatment. This involves the assessment of long term results and potential sequelae. Existing data will be complemented with information about recurrences and complications. The question is: Which treatment method leads to the least numbers of recurrences in the long term with the fewest long term sequelae?

Secondly, the most agreeable, least painful treatment method is to be identified. Therefore we will send out questionnaires to patients that were treated between March 29, 2007 and April 1st, 2008 at the Zurich University Hospital.

ELIGIBILITY:
Inclusion Criteria:

All patients treated during the study period with known address and who did not decease in the meantime.

Exclusion Criteria:

Insufficiently filled out questionnaires; Obvious lack of ability to remember (as tested by control questions); Known mental disability

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients treated between March 29, 2007 and April 1st, 2008 for epistaxis at the ENT Dept. of the Zurich University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 591 (Actual)
Dates: Start 2014-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Number of patients without recurrence | Up to 8 years post-treatment

SECONDARY OUTCOMES:
Discomfort caused by treatment | Up to 1 day post-treatment

OTHER OUTCOMES:
Number of complications due to treatment | Up to 8 years post-treatment
Sequelae due to treatment | Up to 8 years post-treatment

CONTACTS AND LOCATIONS:
Overall Officials: Michael Soyka, Dr.med., Principal Investigator — Zurich University Hospital
Locations (1):
- Zurich University Hospital, Zurich, Canton of Zurich, Switzerland